CLINICAL TRIAL: NCT04892563
Title: Erector Spinae Plane Block for Rib Fracture Analgesia in the Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Dana Sajed, Clinical Associate Professor (Clinican Educator), Emergency Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-21-00066
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Rib Fracture Multiple
MeSH Terms: interventions — Nerve Block; Analgesia; Morphine; Analgesics, Opioid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB Block (Experimental): Patients with rib fracture randomized to block group
  Interventions: Procedure: Erector Spinae Plane Block
- Standard Care (Active Comparator): Patients with rib fracture receiving IV analgesia/standard care
  Interventions: Drug: IV Analgesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Nerve block with local anesthetic in the erector spinae plane
  Other Names: Nerve Block; Erector Spinae Block
  Arms: ESPB Block
Drug: IV Analgesia — IV analgesia, typically Morphine/Opioid medications
  Other Names: Morphine; Opioid
  Arms: Standard Care

SUMMARY:
Rib fractures, while in isolation are self-limited and benign, can be exquisitely painful. Poorly controlled rib fracture pain can compromise respiratory function leading to increased morbidity and mortality, especially in the elderly. Currently, opioid medications are the mainstay of analgesia but are associated with significant adverse effects, such as respiratory depression and delirium. In an effort to improve acute pain in the ED and concomitantly reduce opioid use, ultrasound-guided regional anesthesia has been implemented more frequently The erector spinae plane block (ESPB) is a relatively new ultrasound-guided procedure for thoracic analgesia.

Previously, the serratus anterior plane (SAP) block has been used for this indication. However, typical anatomical distribution limits the effectiveness of the SAP block to anterior rib fractures, while the majority of traumatic rib fractures are posterior, thus require a more central blockade such as the proposed ESPB. The ESPB can be done as a single injection into the superficial structures of the back under ultrasound guidance and as such, is a both a relatively safe and technically easy procedure to perform, especially in comparison to the more traditional alternatives of epidurals, paravertebral and intercostal injections.

There have been no prospective studies evaluating the efficacy and safety of the ESPB in the emergency department setting for acute rib fractures. The investigators hypothesize that the ESPB will provide improved acute pain scores in the emergency department compared to parental analgesia alone. Secondarily, investigators hypothesize that this will translate to less inpatient opioid requirements and improved incentive spirometry values.

DETAILED DESCRIPTION:
Rib fractures, while in isolation are self-limited and benign, can be exquisitely painful. Poorly controlled rib fracture pain can compromise respiratory function leading to increased morbidity and mortality, especially in the elderly. Currently, opioid medications are the mainstay of analgesia but are associated with significant adverse effects, such as respiratory depression and delirium. Additionally, even short courses can predispose to life-long addiction perpetuating the opioid epidemic. In an effort to improve acute pain in the ED and concomitantly reduce opioid use, ultrasound-guided regional anesthesia has been implemented more frequently. As an example, ultrasound-guided peripheral nerve blocks for hip fractures have a promising track record for reducing opioid use and improving pain scores. The erector spinae plane block (ESPB) is a relatively new ultrasound-guided procedure for thoracic analgesia. It was first described in 2016 by Forero, et al., as an effective alternative to traditional neuraxial blockade for post-operative and chronic thoracic pain. A recent literature review by Kot et al., 2019 revealed six prospective studies in post-operative patients concluding that the ESPB was at least as effective as opioids in thoracic pain reduction, easy to use and with a low complication rate. One prospective study in post-operative breast surgery patients demonstrated a reduction in morphine by 65% compared to control. Most literature on the ESPB in the ED are case reports, which demonstrate its versatility in a myriad of clinical situations such as renal colic, acute herpes zoster, acute transverse process fractures, extensive burns, mechanical back pain, acute pancreatitis and acute rib fractures. This review found the ESPB to be effective at reducing pain scores for all reported indications with no complications. The ESPB is a particularly attractive multimodal form of analgesia in the ED where acute traumatic rib fractures are a common presentation. Usually the involuntary splinting from acute pain results in the typical pulmonary complications, but high doses of opioids and the subsequent respiratory depressive effects can lead to higher rates of atelectasis, pneumonia and respiratory failure. In order to combat this "between a rock and a hard place" scenario, regional analgesia has emerged as an effective means of improving both pain respiratory mechanics. Previously, the serratus anterior plane (SAP) block has been used for this indication. However, typical anatomical distribution limits the effectiveness of the SAP block to anterior rib fractures, while the majority of traumatic rib fractures are posterior, thus require a more central blockade such as the proposed ESPB. The ESPB can be done as a single injection into the superficial structures of the back under ultrasound guidance and as such, is a both a relatively safe and technically easy procedure to perform, especially in comparison to the more traditional alternatives of epidurals, paravertebral and intercostal injections. Another consideration of these technically more difficult procedures is that they are relatively contraindicated in the anticoagulated patient precluding a substantial number of elderly patients from their therapeutic benefits. The aforementioned reviews have supported the safety of the ESPB with no complications reported. Specifically, of the 10 case reports utilizing this block in the ED, none reported any complications. The 3 cases reported by Luftig et al, in 2018 specific to ED management of acute rib fractures were technically feasible, highly efficacious and safe. However, there have been no prospective studies evaluating the efficacy and safety of the ESPB in the emergency department setting for acute rib fractures. The investigators hypothesize that the ESPB will provide improved acute pain scores in the emergency department compared to parental analgesia alone. Secondarily, the investigators hypothesize that this will translate to less inpatient opioid requirements and improved incentive spirometry values.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* At least 1 acute rib fracture. Acute defined as within 7 days of presentation.
* Numerical pain score on presentation at least 5 out of 10. This will identify patients that justify the invasive procedure.
* Admitted to hospital for at least 24 hours of observation.
* Be able to consent and participate in study by assuming necessary positioning for intervention

Exclusion Criteria:

* Hypotension/shock (shock index >1.0, SBP < 90)
* Distracting injury not amenable to ESPB as determined by the enrolling physician. (i.e extremity fracture, burn, laceration, contusion, joint dislocation, etc.)
* Examples of patients not able to consent/participate are intubated patients or patients in spinal precautions (i.e c-collar)
* Known hypersensitivity to local anesthetic
* Evidence of infection at the proposed site of injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
To determine the effectiveness of the ESPB for pain management of acute rib fractures in the emergency department using a 10 point isual analog scale | 0, 1, 2 and 24 hours assessment
  Change in pain level from fractures as measured using a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mailhot, MD, Principal Investigator — LAC+USC Medical Center

IPD SHARING:
Plan to Share IPD: No